CLINICAL TRIAL: NCT06550596
Title: A Randomized Controlled Multicenter Clinical Trial Evaluating Dehydrated Human Amnion Membrane (dhAM) and Standard of Care Versus Standard of Care Alone in Nonhealing Diabetic Foot Ulcers
Brief Title: Dehydrated Human Amnion Membrane and Standard of Care Versus Standard of Care Alone in Nonhealing Diabetic Foot Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Axolotl Biologix (Industry)
Collaborators: SerenaGroup, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AXOLCAMP
Record Dates: First submitted 2024-08-05; First posted 2024-08-13 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Foot; Ulcer Foot; Foot Ulcer; Diabetic Foot Ulcer
Keywords: Cellular, Acellular, Matrix-like Product (CAMP); Dehydrated Human Amnion Membrane (dhAM); Vascular Diseases; Leg Ulcer; Ulcer leg; Skin Ulcer; Diabetes Complications; Diabetes Mellitus; Diabetic Neuropathies; Foot Diseases; Diabetic Foot; Foot Ulcer; Ulcer
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer; Vascular Diseases; Leg Ulcer; Skin Ulcer; Diabetes Complications; Diabetes Mellitus; Diabetic Neuropathies; Foot Diseases; Ulcer | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: AXOLCAMP is a multi-center, open label, randomized controlled trial to determine the efficacy of dhAM plus SOC versus SOC alone in achieving complete closure of nonhealing diabetic foot ulcers.
  over 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Standard of care will be cleaning, debridement, ulcer moisture balance, and offloading.
  Interventions: Other: Standard of Care
- Axolotl DualGraft + SOC (Experimental): Axolotl DualGraft is a dehydrated human amnion membrane.
  Interventions: Other: Axolotl DualGraft + SOC

INTERVENTIONS:
Other: Standard of Care — Beginning at the screening visit, participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Standard of Care
Other: Axolotl DualGraft + SOC — Participants will receive weekly applications of Axolotl DualGraft and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Axolotl DualGraft + SOC

SUMMARY:
The purpose of this study is to evaluate the efficacy of dehydrated human amnion membrane (dhAM) and standard of care (SOC) versus SOC alone in the closure of nonhealing diabetic foot ulcers (DFUs).

DETAILED DESCRIPTION:
AXOCAMP is a multi-center randomized controlled clinical trial. The study will evaluate the efficacy of dehydrated human amnion membrane (dhAM) and standard of care (SOC) versus SOC alone in the closure of nonhealing diabetic foot ulcers (DFUs).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age or older.
* Subjects must have a diagnosis of type 1 or 2 Diabetes mellitus.
* At randomization subjects must have a target ulcer with a minimum surface area of 1.0 cm2 and a maximum surface area of 5.0 cm2 measured post debridement.
* The target ulcer must have been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care prior to the initial screening visit.
* The target ulcer must be located on the foot with at least 50% of the ulcer below the malleolus.
* The target ulcer must be Wagner 1 or 2 grade, extending at least through the dermis or subcutaneous tissue and may involve the muscle provided it is below the medial aspect of the malleolus. The ulcer may not include exposed tendon or bone.
* The affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

  1. ABI ≥ 0.7 and ≤ 1.3;
  2. TBI ≥ 0.6;
  3. TCOM ≥ 40 mmHg;
  4. PVR: biphasic.
* If the subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
* The subject must consent to using the prescribed offloading method for the duration of the study.
* The subject must agree to attend the weekly study visits required by the protocol.
* The subject must be willing and able to participate in the informed consent process.

Exclusion Criteria:

* A subject known to have a life expectancy of < 6 months is excluded.
* The subject is excluded if the target ulcer is not secondary to diabetes.
* If the target ulcer is infected or if there is cellulitis in the surrounding skin, the subject is excluded.
* If there is evidence of osteomyelitis complicating the target ulcer, the subject is excluded.
* A potential subject cannot have an infection in the target ulcer or in a remote location that requires systemic antibiotic therapy.
* A subject receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of Prednisone per day or equivalent) or cytotoxic chemotherapy is excluded.
* The topical application of steroids to the ulcer surface within one month of initial screening is not permitted.
* A subject with a previous partial amputation on the affected foot is excluded if the resulting deformity impedes proper offloading of the target ulcer.
* The subject is excluded if the surface area of the target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit ("historical" run-in period). Photographic planimetry is not required for measurements taken during the historical run-in period (e.g. calculating surface area using length x width is acceptable).
* The subject is excluded if the surface area measurement of the Target ulcer decreases by 20% or more during the 2-week screening phase: the 2 weeks from the initial screening visit (S1) to the TV-1/randomization visit, during which time the subject received SOC.
* A subject is excluded if they are malnourished: a score of less than 17 on the Mini Nutritional Assessment (MNA).
* A Subject with an acute Charcot foot, or an inactive Charcot foot, that impedes proper offloading of the target ulcer is excluded.
* Women who are pregnant or considering becoming pregnant within the next 6 months are excluded.
* A potential subject with end stage renal disease requiring dialysis is excluded.
* A subject who, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments is excluded.
* A Subject treated with hyperbaric oxygen therapy or a Cellular Acellular, or Matrix-like Product (CAMP) in the 30 days prior to the initial screening visit is excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy of dhAM + SOC vs SOC | 1-12 Weeks
  To determine the efficacy of dhAM plus SOC versus SOC alone in achieving complete closure of nonhealing diabetic foot ulcers over 12 weeks.

SECONDARY OUTCOMES:
Time to closure for the target ulcer | 1-12 weeks
  To determine the proportion of ulcers that heal over 12 weeks for dhAM plus SOC versus SOC alone (Time to closure).
Percent area reduction | 1-12 weeks
  To determine the percent area reduction (PAR) of the ulcer over the 12-week treatment period.
Adverse events | 1-12 Weeks
  To demonstrate a reduction in adverse events in subjects receiving dhAM plus SOC versus SOC alone.
Determine improvement in quality of life using Wound Quality of Life questionnaire | 1-12 weeks
  Quality of Life is assessed using the Wound Quality of Life (wQOL) checklist at TV1, TV3, TV7, TV11, and TV12. This assessment will be used to compare patients receiving dhAM + SOC vs SOC.
Determine improvement in quality of life using Forgotten Wound Score questionnaire | 1-12 weeks
  Quality of life is assessed using the Forgotten Wound Score (FWS) at TV1, TV3, TV7, TV11, and TV12. This assessment will be used to compare patients receiving dhAM + SOC vs SOC.

OTHER OUTCOMES:
Proportion of ulcers that heal in patients 65 years and older | 1-12 weeks
  To determine the proportion of ulcers that heal in patients 65 years or older for dhAM plus SOC versus SOC alone.
Determine the effect of chronic inhibitory bacterial load (CIBL) on wound closure | 1-12 weeks
  To determine the effect of chronic inhibitory bacterial load (CIBL) as assessed by fluorescence imaging on wound closure. Fluorescent imaging will be assessed at TV1, TV4, TV8, and TV12.

CONTACTS AND LOCATIONS:
Locations (1):
- Performance Foot and Ankle Specialists, Thousand Oaks, California, United States

IPD SHARING:
Plan to Share IPD: No